CLINICAL TRIAL: NCT02895425
Title: Réseau, Epidémiologie, Information, Néphrologie (Network Epidemiology Information Nephrology)
Brief Title: Registry for End Stage Renal Failure
Acronym: REIN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier de Cayenne (Other)
Responsible Party: Sponsor
Other Study IDs: REIN
Record Dates: First submitted 2016-09-06; First posted 2016-09-09 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-09

CONDITIONS: End Stage Renal Failure
Keywords: Renal Transplant
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Registries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Registry (No intervention)

SUMMARY:
The rein registry collects case record data from patients with end stage renal disease followed in French Guiana. This allows to generate incidence and rates for terminal renal disease, mortality rates for each territory. The regional data are pooled in order to get national statistics for end stage renal disease and transplantation activity in order to adapt prevention to the main causes of renal failure and treatment and care infrastructure.

ELIGIBILITY:
Inclusion Criteria:

* End Stage Renal Failure

Exclusion Criteria:

* Refusal to participate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient with End Stage Renal Failure followed in one of the dialisys sites in frnech Guiana
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-01 (Actual); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Death | 10 years
Transplant | 10 years

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital of Cayenne, Cayenne, French Guiana, France

IPD SHARING:
Plan to Share IPD: No